CLINICAL TRIAL: NCT04910191
Title: Collecting Respiratory Sound Samples From Corona Patients to Extend the Diagnostic Capability of VOQX Electronic Stethoscope to Diagnose COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanolla (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: VOQX
Record Dates: First submitted 2021-02-23; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: COVID-19; Diagnostic; Viral infection disease; Electronic stethoscope
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): Up to 200 patients will participate in this open study. Before each examination with the study device, data from each patient (Current medical condition, medical history and demographic data) will be inserted to a computer and added to the database of the study for further processing in conjunction with the study device results.
  The study device electronic stethoscope membrane will be put on the patient's chest area in predefined anterior and posterior points. At the end of each examination the data will be transferred to a computer and stored in the patient's file. Each patient will be requested to attend the examination once.
  Interventions: Diagnostic Test: Electronic stethoscope

INTERVENTIONS:
Diagnostic Test: Electronic stethoscope — Electronic stethoscope
  Other Names: VOQX

SUMMARY:
Technological developments in the recent decades has enabled the integration of electronic and digital components in the stethoscope design, in an attempt to improve auditory performance and, moreover, to assist in improving user's diagnostic accuracy by incorporating computerized, digital technologies, artificial intelligence capabilities and deep-learning-based algorithms enhancing these devices.

We believe that these technologies can be used to significantly improve the diagnostic performance in the primary care phase, by means of a sophisticated stethoscope that enables auscultation to sounds and signals typically found in the sub-sound frequency level. Their transformation into the sound range, and the use of artificial intelligence and machine learning techniques to characterize sound patterns that correspond to specific problems or diseases can substantially enhance the physician's or other care giver's performance to the benefit of the patients.

At this stage, the software in development does not purport to make diagnostic decisions, but only to provide information that will enhance decision and diagnosis making process, therefore enable a more accurate and definitive diagnostic decision and perhaps decrease the number of additional diagnostic tests requested.

DETAILED DESCRIPTION:
Up to 200 patients will participate in an open, prospective and multi-center study.

Patients diagnosed as positive to COVID-19 will be referred to a VOQX examination. All patients will receive detailed explanation about the purpose of the examination, its impact and will provide their consent prior to the examination. The VOQX device output will have no influence on the decision-making process of the physicians and care givers. The VOQX Stethoscope membrane will be put on the patient's chest area in predefined anterior and posterior points. The data collected in the form of breath sound signals in particular infra-sound will be transferred to an external computer and processed by machine learning algorithm developed by the company. The algorithm will seek patterns typical for the diagnosed disease for each corresponding case diagnosed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years
* RT-PCR positive for COVID 19
* Patients diagnosed with the following pulmonary pathology:

  * Pneumonia
  * Pulmonary edema
  * Bronchitis
  * Acute asthmatic attack
  * Emphysema
  * Or Normal (e.g. asymptomatic patients)
* The diagnosis is confirmed if possible, by:

  * Anamnesis
  * Physical examination
  * X-ray
  * Suggestive blood test - CBC
  * Pulse oximetry

Exclusion Criteria:

* Pregnant women
* Chest malformation
* Unconsciousness
* Subject that need a guardian
* Weigh above 150 Kg.
* Patients with current shortness of breath
* Patients currently assisted by breathing machine such as CPAP or other

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Performance outcome | Through study completion, an average of 1 year
  Detection and identification of pulmonary sound signals ranging from infra-sound to auditory sound which are typical to specific pathologies of COVID-19
Performance outcome | through study completion, an average of 1 year
  Use machine learning technologies to identify the above sound patterns and corresponding pathologies

CONTACTS AND LOCATIONS:
Overall Officials: David Linhard, Study Director — Sanolla
Locations (3):
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Hille Yaffe Medical Center, Hadera
  - Shamir Medical Center (Assaf Harofah), Zrifin